CLINICAL TRIAL: NCT04492930
Title: The Effect of 14:10 Hour Time Restricted Eating on Body Weight and Metabolic Markers: An 8-Week Pilot Study in Individuals With Obesity
Brief Title: Effect of 14:10 Time-Restricted Eating on Body Weight and Metabolic Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jenny Craig, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRM-102
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Time Restricted Feeding
Keywords: body weight; weight loss; ketones; blood glucose
MeSH Terms: conditions — Intermittent Fasting; Body Weight; Weight Loss; Ketosis | interventions — Clinical Protocols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator (Active Comparator): Time restricted eating
  Interventions: Behavioral: 12:12 Regimen
- Intervention (Experimental): Time restricted eating
  Interventions: Behavioral: 14:10 Regimen

INTERVENTIONS:
Behavioral: 14:10 Regimen — 14 hours of fasting, followed by a 10-h diet regimen that includes a fasting snack at 12 hours from the start of the fasting period
  Arms: Intervention
Behavioral: 12:12 Regimen — 12 hours of fasting, followed by a 12-h diet regimen
  Arms: Comparator

SUMMARY:
The purpose of this study is to investigate the effect of engaging in time restricted eating schedule on body weight, blood glucose, and ketones (breath acetone) in individuals with obesity.

DETAILED DESCRIPTION:
There are significant metabolic and weight reduction benefits associated with time restricted feeding/eating. Time restricted eating splits the day into a period of regeneration (non-eating or natural fasting) and a period of nourishing. Providing the body a period of regeneration allows the body to go into ketosis, or the elevation in circulating ketone bodies, a byproduct of fat metabolism. Breath acetone concentration is a good predictor of ketosis and loss of body fat. In healthy individuals, low concentrations of breath acetone are 1 to 2 ppm. Engaging in weight loss via nutritional ketosis (engaging in high-fat, low-carbohydrate diets, caloric restriction diets, or fasting) increases fat utilization, resulting in increased formation of ketone bodies and breath acetone concentrations ranging from 4 to 30 ppm. In individuals with obesity, nutritional ketosis facilitates weight loss and improves insulin sensitivity, lipid profile, and reduces inflammatory markers.

This study will investigate the effect of participating in two different time restricted eating schedules for 8 weeks on body weight, blood glucose, and ketones.

After being informed about the study and potential risks, all eligible participants giving written informed consent will be randomized to a different time restricted eating schedule (ie, one group fasts for a longer period of time). In both of these groups, fasting will begin each evening and end the following morning.

This is a remote study. All procedures will be conducted at home.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female individuals between the age of 18 to 65 years (inclusive) at the time of signing the informed consent
2. Enrollment in the Jenny Craig® Rapid Results™ program
3. Access to a tablet or smartphone with a camera and internet access
4. Body mass index (BMI) at least 30 kg/m2
5. Ability to use a glucometer and Levl device (measures breath acetone)
6. Female participants of childbearing potential will agree to avoid pregnancy during the study. Medically acceptable methods of contraception include oral contraceptive medication, an intrauterine device (IUD), an implantable contraceptive (such as Implanon), an injectable contraceptive (such as Depo-Provera), a barrier method (such as condom or diaphragm with spermicide), abstinence, or having exclusive sexual relations with a vasectomized or same sex partner.
7. Capable of giving signed informed consent.

Exclusion Criteria:

1. Current use of the medications indicated for weight management or treatment of diabetes or for treatment of psychosis
2. Serious allergy to corn, corn products, or gluten (due to the number of Jenny's Cuisine® items that contain these food ingredients) that results in throat swelling, rash, hives, or anaphylactic shock
3. Serious allergy to milk, soy, wheat, peanuts, or tree nuts that results in throat swelling, rash, hives, or anaphylactic shock
4. Celiac disease
5. Currently being treated with hemodialysis
6. Currently being treated for anorexia/bulimia
7. Require a special diet (vegan, kosher, or halal)
8. Had a baby within the last 6 weeks
9. Are currently breastfeeding
10. Are pregnant
11. Bariatric surgery within the previous 3 years
12. Individuals belonging to the following vulnerable populations (people with disabilities, people who cannot read, educationally disadvantaged, individuals with a serious or life threatening illness, prisoners, non-English speakers, economically disadvantaged individuals, employees of the study sponsor)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Week 4
  Change from baseline body weight in the intervention group
Change in ketone levels (breath acetone) | Week 8
  Change from baseline in breath acetone in the intervention group
Change in blood glucose | Week 8
  Change from baseline in blood glucose in the intervention group

SECONDARY OUTCOMES:
Change in body weight | Week 8
  Change from baseline body weight in the intervention group
Difference in weight loss between groups | Weeks 4 and 8
  Difference in the change from baseline in body weight between the intervention and control groups
Time to first meal | Weeks 4 and 8
  Change from baseline in the length of time from consumption of the fasting snack until initiation of the first meal in the intervention group

OTHER OUTCOMES:
Correlation between weight loss and change in ketone levels (breath acetone) | Week 8
  Correlation between the change from baseline in breath acetone and the change from baseline in body weight

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Peeke, MD, Study Director — Jenny Craig, Inc.
Locations (1):
- Jenny Craig, Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized dataset of selected variables that underlie results in a publication. Some data may not be amenable to complete anonymization and will not be shared to ensure appropriate confidentiality of participant's data.
Supporting Information: Study Protocol
Time Frame: beginning 6 months after publication
Access Criteria: Upon appropriate data request by other scientists